CLINICAL TRIAL: NCT02534077
Title: Compassionate Use of an Intravenous Fat Emulsion Comprised of Fish Oil in the Treatment of Parenteral Nutrition Induced Liver Injury in Infants
Brief Title: Intravenous Fat Emulsion Comprised of Fish Oil in the Treatment of Parenteral Nutrition Induced Liver Injury in Infants
Status: Approved for marketing | Type: Expanded Access
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: WIRB Study# 1155515
Record Dates: First submitted 2015-07-27; First posted 2015-08-27 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2019-04

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis
Keywords: omegaven; cholestasis; parenteral nutrition associated liver disease
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

INTERVENTIONS:
Dietary Supplement: Omegaven — Therapy with Omegaven will be provided at a dose of 1 gm/kg/day (by continuous infusion). Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition.
  Other Names: omega-3 enriched fat emulsion
Drug: Omegaven — Treatment will be given for as long as the child needs any TPN AND has a conjugated bilirubin greater than 2 mg/dL for a maximum of 2 years.
Drug: Omegaven — If the bilirubin is less than 2 mg/dL but the child still requires TPN, then the Omegaven will be continued until the infant no longer requires TPN.

SUMMARY:
To provide a mechanism for critically ill infants with parenteral nutrition (PN) associated cholestasis to receive Omegaven for compassionate use situations for which there are no satisfactory alternative treatments.

DETAILED DESCRIPTION:
Compassionate Use

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill infants with either a known anatomic short gut (greater than 50% of the bowel removed) or known severe dysmotility of the gut reflecting non-functional gut similar to anatomic short gut will be offered Omegaven® when their direct bilirubin reaches 2 mg/dL. Infants who do not meet the above criteria for anatomic or dysfunctional short gut will be allowed to receive Omegaven® when their direct bilirubin reaches 4 mg/dL. The qualifying measurements of 2 mg/dL or 4 mg/dL direct bilirubin must be consecutive and obtained at least 24 hours apart.
2. Be expected to require intravenous nutrition for at least an additional 28 days
3. Patient must have documented failure of or ineligibility for the following therapies to prevent progression of PNALD:

   * Reduction of Intralipid® to 1 g/kg/day
   * Limiting trace minerals including copper and manganese
   * Initiation and use of Ursodiol
   * Cycling of parenteral nutrition
   * Advancement of enteral feedings
4. Parental informed consent must be signed.

Exclusion Criteria:

1. Have a congenitally lethal condition (e.g. Trisomy 13).
2. Have clinically severe bleeding not able to be managed with routine measures.
3. Have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
4. Have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves.
5. Has culture positive sepsis

Ages: 14 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Kaashif Ahmad, MD, Principal Investigator — Pediatrix
Locations (1):
- Children's Hospital of San Antonio, San Antonio, Texas, United States